CLINICAL TRIAL: NCT00030563
Title: A Phase II Study Of Adjuvant Intravenous Irinotecan Following Resection With Or Without Radiofrequency Ablation (RFA), Of Hepatic Metastases From Colorectal Carcinoma
Brief Title: Surgery With or Without Radiofrequency Ablation Followed by Irinotecan in Treating Patients With Colorectal Cancer That is Metastatic to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raymond Yeung, Professor, Division of General Surgery, Oncology, University of Washington
Purpose: Treatment
Other Study IDs: 18033; UWASH-1200; CWRU-040106; UWASH-440E-ONC-0020-250; NCI-G01-2045; CWRU-UWMC-1200
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Chemotherapy, Adjuvant; Radiofrequency Ablation

INTERVENTIONS:
Drug: irinotecan hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses high-frequency electric current to kill tumor cells. Combining radiofrequency ablation with surgery may kill more tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug after surgery and radiofrequency ablation may kill any remaining tumor cells.

PURPOSE: Phase II trial to determine the effectiveness of surgery with or without radiofrequency ablation followed by irinotecan in treating patients who have colorectal cancer that is metastatic to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the disease-free survival in patients with hepatic metastases from primary colorectal carcinoma treated with surgical resection with or without radiofrequency ablation followed by irinotecan.
* Determine the overall survival in patients treated with this regimen.
* Determine the treatment-related toxicity of this regimen in these patients.
* Correlate the measurement of molecular markers with clinical outcome in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment with radiofrequency ablation in addition to resection (yes vs no).

Patients undergo surgical resection with or without radiofrequency ablation. Beginning 4-8 weeks after surgery, patients receive irinotecan IV over 90 minutes on day 1. Chemotherapy repeats every 3 weeks for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary colorectal adenocarcinoma
* Hepatic metastases that are considered completely resectable

  * No more than 4 metastases by dual phase CT scan OR
* Hepatic metastases that are not completely resectable but are amenable to complete destruction with resection and radiofrequency ablation

  * More than 4 metastases allowed if all disease can be resected or destroyed in situ with radiofrequency ablation
* No extrahepatic disease in any location
* No recurrent or second primary colorectal cancer by colonoscopy within the past year
* Received prior adjuvant chemotherapy with a fluorouracil-based regimen with the last dose at least 1 month prior to surgery
* No prior radiofrequency ablation with residual viable intrahepatic disease by CT scan
* No plans to be treated with radiofrequency ablation alone without surgical resection

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 5 times ULN
* No Gilbert's disease or other known defect in hepatic conjugation or glucuronidation

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure requiring therapy

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 30 days after study
* No other malignancy within the past 5 years except inactive non-melanoma skin cancer or carcinoma in situ of the cervix
* No active serious infection
* No other serious underlying medical condition or severe concurrent disease that would preclude study participation
* No dementia, significantly altered mental status, or psychiatric illness that would preclude study participation
* No known hypersensitivity to irinotecan
* No known infection with HIV or AIDS
* No uncontrolled diabetes mellitus
* No history of seizures
* No drug or alcohol abuse within the past year

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior irinotecan

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to more than 30% of bone marrow
* No prior radiotherapy to the liver
* At least 3 months since prior radiotherapy to the pelvis or other areas

Surgery:

* See Disease Characteristics
* No prior resection of hepatic metastases (wedge biopsy allowed)

Other:

* No concurrent phenytoin, phenobarbital, or other antiepileptic medication
* No concurrent enrollment in other investigational drug trials

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2004-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G. Billingsley, MD, Study Chair — University of Washington
Locations (3):
- United States (2):
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Washington School of Medicine, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada